CLINICAL TRIAL: NCT05154045
Title: Postprandial Glycemic Response to a Diabetes-Specific Formula and Oatmeal in Individuals With Type 2 Diabetes
Brief Title: Postprandial Glycemic Response in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BL61
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Formula (Experimental): One 330 ml serving of study product
  Interventions: Other: Experimental Formula
- Test Meal (Active Comparator): 40 g Instant oatmeal
  Interventions: Other: Test Meal

INTERVENTIONS:
Other: Experimental Formula — Diabetes-specific study formula
  Arms: Experimental Formula
Other: Test Meal — Instant oatmeal
  Arms: Test Meal

SUMMARY:
This is a randomized, controlled, crossover study to compare the effects of two treatments on postprandial glucose in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 and ≤ 75 years.
* Participant has type 2 diabetes as evidenced by use of oral antihyperglycemic medication(s) with constant dose for at least two months prior to screening and baseline visit. Participant is able to maintain medication number, type and dose throughout the duration of study.
* Participant with a BMI > 18.5 and ≤ 40.0 kg/m2
* Participant is weight stable for the two months prior to the screening visit.
* Male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
* If the participant is on a chronic medication such as an anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, the dosage must be constant for at least two months prior to screening and baseline visit. Participant is able to maintain medication number, type and dose throughout the duration of study.
* Participant is willing to follow protocol as described, including consumption of study product per protocol and completing any forms needed throughout the study.
* Participant has at least a two-week washout period between completion of a previous research study that required ingestion of any study food or drug and Visit 2 when assigned study product is consumed.
* Participant is willing to refrain from taking non-study diabetes-specific formulas over the entire course of the study.
* Participant has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

* Participant has a screening HbA1c level < 7% or ≥ 10%.
* Participant uses exogenous insulin or GLP-1 agonists or DPP-4 inhibitors for glucose control.
* Participant has confirmed type 1 diabetes and/or had history of diabetic ketoacidosis.
* Participant has current infection, inpatient surgery or received systemic corticosteroid treatment in the last 3 months; or received antibiotics in the last 3 weeks.
* Participant has active malignancy.
* Participant has significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure.
* Participant has end stage organ failure or was post organ transplant.
* Participant has a history of renal disease or severe gastroparesis.
* Participant has current hepatic disease.
* Participant has had bariatric surgery including gastric balloon; history of gastrointestinal disease or intestinal surgery that can interfere with consumption or digestion or absorption of study product.
* Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV.
* Participant has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures.
* Participant is taking any herbals, dietary supplements, or medications, other than allowed anti-hyperglycemic medications, during the past four weeks prior to screening visit that could profoundly affect blood glucose or appetite.
* Participant uses diabetes-specific formula(s), defined as more than one eating occasion per week in the last three months.
* Participant has clotting or bleeding disorders. The use of Plavix® or a similar anticoagulant drug with no reported difficulty during blood draws is allowed and participant is able to maintain medication number, type and dose throughout the duration of study.
* Participant participates in another study that has not been approved as a concomitant study by AN.
* Participant has an allergy or intolerance to any ingredient in the study product, as reported by the participant.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Glucose positive area under the curve (AUC) | 0 to 240 minutes
  Calculated from blood samples

SECONDARY OUTCOMES:
Insulin positive area under the curve (AUC) | 0 to 240 minutes
  Calculated from blood samples
Insulin peak value | 0 to 240 minutes
  Calculated from blood samples
Glucose peak value | 0 to 240 minutes
  Calculated from blood samples
Insulin peak time | 0 to 240 minutes
  Calculated from blood samples
Glucose peak time | 0 to 240 minutes
  Calculated from blood samples
Insulin Concentrations | 0 to 240 minutes
  Calculated from blood samples
Glucose Concentrations | 0 to 240 minutes
  Calculated from blood samples

OTHER OUTCOMES:
Glucagon-Like Peptide-1 (GLP-1) positive area under the curve (AUC) | 0 to 240 minutes
  Calculated from blood samples
Glucagon-Like Peptide-1 (GLP-1) peak value | 0 to 240 minutes
  Calculated from blood samples
Glucagon-Like Peptide-1 (GLP-1) peak time | 0 to 240 minutes
  Calculated from blood samples
Glucagon-Like Peptide-1 (GLP-1) Concentrations | 0 to 240 minutes
  Calculated from blood samples
Appetite Questionnaire | Study Day 1 to Study Day 7
  5 Visual analog scales; Including Score from Not at All to Extremely or Nothing to Most
Sensory Questionnaire | Study Day 1 to Study Day 7
  10 sensory and hedonic questions; Up to 9-Point Likert Scale questions including Dislike Extremely to Like Extremely or Much too to Much less or Not at all to Extremely

CONTACTS AND LOCATIONS:
Overall Officials: Sara Thomas, PhD, RDN, Study Chair — Abbott Nutrition
Locations (3):
- United States (3):
  - Finlay Medical Research 3322, Greenacres City, Florida
  - Finlay Medical Research 3323, Miami, Florida
  - Great Lakes Clinical Trials, LLC, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No